CLINICAL TRIAL: NCT02299544
Title: Safety and Performance of the BlueWind System for the Treatment of Patients With Overactive Bladder (OAB) Amended to Allow Extended Follow up of the Patients
Brief Title: BlueWind Medical System for the Treatment of Patients With OAB
Acronym: OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BlueWind Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-03-001
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2018-11

CONDITIONS: Over Active Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OAB (Experimental): Patients with overactive bladder (OAB) with or without urge incontinence.
  Two patient populations will be enrolled in the study:
  Patients with no previous treatment with percutaneous tibial nerve stimulation (PTNS) [de novo patient group] and Patients with a documented success on PTNS therapy [prior-PTNS group]. Documented success on PTNS is defined by a ≥50% reduction in urinary frequency, and/or ≥50% fewer incontinence episodes, or a return to normal voiding frequency [<8 voids/day], based on retrospective diary review.
  All patients will be treated with BlueWind Medical System.
  Interventions: Device: BlueWind Medical system

INTERVENTIONS:
Device: BlueWind Medical system — The BlueWind Medical System is intended for the treatment of patients with overactive bladder (OAB) including urinary urgency frequency and urge incontinence.

SUMMARY:
BlueWind system safety and performance in treatment of patients diagnosed with overactive bladder (OAB)

DETAILED DESCRIPTION:
BlueWind Medical system safety and performance in treatment of patients diagnosed with overactive bladder (OAB)

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Male or female aged 18 - 80.
* Patient agrees to attend all follow-up evaluations and is willing to completely and accurately fill out voiding diaries and questionnaires, and is willing to complete required exams and tests.
* Patients with overactive bladder symptoms:
* Urinary frequency greater than 8 times/24 hours AND/OR Urinary urgency leaks of at least 2 leaks on 3 day voiding diary
* Patient who has failed conservative treatment after at least 6 months of treatment
* Patients with normally functioning upper urinary tract.
* Patients with no clinical evidence of a neurological S2-S4 motor sensory deficit.
* Prior PTNS Group: Patients who have had successful PTNS treatment (successful treatment is defined as ≥50% reduction in urinary frequency, and/or ≥50% fewer incontinence episodes, or a return to normal voiding frequency [<8 voids/day], based on retrospective diary review).
* De novo Patient Group: Patient who passes the BlueWind compatibility test.

Exclusion Criteria:

* Any metal implant in the area of BlueWind Medical implantation site.
* Patients who have not had stable OAB medications for at least 30 days.
* Patients who have received botulinum toxin injections within the past 6 months.
* Previous urinary incontinence surgery or implantation of artificial graft material within the last 6 months.
* Any spinal or genitourinary surgery within the last 6 months. Pelvic pain disorders
* Obvious clinically demonstrated genuine stress incontinence.
* Any neurological disease or disorder including neuropathy or injury resulting in neuropathy.
* Current urinary tract infection, presence of urinary stone and/or urinary tract malignancy (i.e. tumor, vesicourethral reflux, etc.)
* Pelvic radiotherapy and chemotherapy.
* Severe uncontrolled diabetes.
* Patients anticipating magnetic resonance imaging (MRI) exams.
* Presence of cystocele, enterocele or rectocele of grade 3 or 4.
* Prior PTNS Group: Patients who are receiving concomitant nerve stimulation therapies for OAB treatment, except for PTNS maintenance therapy.
* De novo Patient Group: Patients who have received or are receiving nerve stimulation therapies for OAB treatment, including PTNS.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02; Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events | 6 months
  Incidence of serious adverse events system and or procedure related
Incidence of serious adverse events (amended) | 36 months
  Incidence of serious adverse events system and or procedure related (amended)

CONTACTS AND LOCATIONS:
Overall Officials: John Heesakkers, MD, Principal Investigator — Principal Investigator
Locations (6):
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven
  - Maastricht UMC, Maastricht
  - Radboud university medical center Department of Urology, Nijmegen
- United Kingdom (3):
  - Southmead Hosital, Bristol
  - College Hospital and National Hospital for Neurology and Neurosurgery, London
  - St. Mary's Hospital, Imperial College, London